CLINICAL TRIAL: NCT06717477
Title: Streamlining Care for Patients With Compression Neuropathies: The Carpal Tunnel Plus Pathway
Acronym: CTS+ Pathway
Status: Enrolling by invitation | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kristine Chapman, Clinical Professor, University of British Columbia
Other Study IDs: H24-03066
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Carpal Tunnel Syndrome; Patient Satisfaction; Care Pathway
MeSH Terms: conditions — Carpal Tunnel Syndrome; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective (Pre-Intervention): Participants in this arm were treated for carpal tunnel syndrome before the Carpal Tunnel Plus Pathway was implemented.
- Prospective (Post-Intervention): Participants in this arm were treated for carpal tunnel syndrome after the Carpal Tunnel Plus Pathway was implemented.
  Interventions: Procedure: Changes to the care pathway for carpal tunnel syndrome (The Carpal Tunnel Plus Pathway)

INTERVENTIONS:
Procedure: Changes to the care pathway for carpal tunnel syndrome (The Carpal Tunnel Plus Pathway) — Changes to the care pathway for carpal tunnel syndrome. Features of the CTS+ pathway include new referral form, care map for mild, moderate and severe CTS established, point or care ultrasound with steroid injection introduced, and expedited referral to surgeons.
  Groups: Prospective (Post-Intervention)

SUMMARY:
The goal of this clinical trial is to assess the impact of a new care pathway (the Carpal Tunnel Plus Pathway) in patients with carpal tunnel syndrome. The main questions it aims to answer are:

1. What was the effect of the Carpal Tunnel Plus Pathway on wait times between each step of the care pathway (e.g. from referral to initial consult, from initial consult to surgical consult, etc.)?
2. How satisfied are patients with the care they received through the Carpal Tunnel Plus Pathway?

Researchers will compare wait times pre- and post- Pathway implementation to see if there was any change.

Participants will be asked to complete a short patient satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Referred to the Vancouver General Hospital Neuromuscular Disease Unit or St. Paul's Hospital with a confirmed diagnosis of carpal tunnel syndrome
* Ability to understand English

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective: Patients age 18 or over seen by study surgeons for CTS. Prospective: patients age 18 or over with carpal tunnel syndrome seen at SPH or Vancouver Hospital EMG lab.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Wait times | From initial referral to surgery/injection (variable, but approximately 9 months)
  Time between each step of the care pathway (e.g. from referral to EMG/neurologic consultation, from referral to surgical consultation, from surgical consultation to surgery)
Patient satisfaction | Immediately after surgery/injection appointment
  Patients will be asked to complete a short questionnaire to indicate their level of satisfaction with the care that they received. The custom survey will consist of 4 questions on various aspects of their care that participants will rate on a scale of 1-5 (1 = not at all satisfied, 5 = very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Chapman, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Only group averages/summary measures will be included in any publications.

REFERENCES:
- See also: Website for the Carpal Tunnel Plus Pathway — https://www.vancouverneuromuscular.ca/carpal-tunnel-plus-clinic